CLINICAL TRIAL: NCT02806765
Title: Effects of a Single Nutrient Supplementation on Dynamic Stability in Community Dwelling Older Adults
Brief Title: Effect of Dietary Supplementation on Dynamic Stability
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Screened 34 participants and only 3 participants met the inclusion criteria, the study was stopped and screening data will be analyzed for associations.
Sponsor: Arizona State University (Other)
Collaborators: Abbott Nutrition (Industry); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Thurmon E. Lockhart, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ANAM1308
Record Dates: First submitted 2016-06-07; First posted 2016-06-21 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Aging
Keywords: Dynamic Stability; Postural Stability; Gait Speed; Hand Grip Strength; Timed Get-up and Go; Older Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement (Experimental): This experimental arm reflects administration of a softgel capsule containing a dose of (1S,3Z)-3-[(2E)-2-[(1R,3aS,7aR)-7a-methyl-1-[(2R)-6-methylheptan-2-yl]-2,3,3a,5,6,7-hexahydro-1H-inden-4-ylidene]ethylidene]-4-methylidenecyclohexan-1-ol below the upper tolerable limit
  Interventions: Dietary Supplement: (1S,3Z)-3-[(2E)-2-[(1R,3aS,7aR)-7a-methyl-1-[(2R)-6-methylheptan-2-yl]-2,3,3a,5,6,7-hexahydro-1H-inden-4-ylidene]ethylidene]-4-methylidenecyclohexan-1-ol
- Control (Experimental): This experimental arm reflects administration of placebo in softgel capsule
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: (1S,3Z)-3-[(2E)-2-[(1R,3aS,7aR)-7a-methyl-1-[(2R)-6-methylheptan-2-yl]-2,3,3a,5,6,7-hexahydro-1H-inden-4-ylidene]ethylidene]-4-methylidenecyclohexan-1-ol — 25 micrograms of (1S,3Z)-3-[(2E)-2-[(1R,3aS,7aR)-7a-methyl-1-[(2R)-6-methylheptan-2-yl]-2,3,3a,5,6,7-hexahydro-1H-inden-4-ylidene]ethylidene]-4-methylidenecyclohexan-1-ol every day for 6 months
  Arms: Dietary Supplement
Other: Control — Placebo in Softgel form
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether specific nutrient supplementation can improve dynamic stability in older adults.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of a single nutrient dietary supplement on dynamic stability in an older population. Dynamic stability, or walking stability, will be assessed with accelerometers while subjects are walking on a flat surface for about 60 seconds. Dynamic stability will be defined by the maximum Lyapunov exponent (maxLE), Floquet multiplier, or motor control timing, change from baseline. Postural stability will also be measured in a still and standing subject, with foot placement standardized on a force plate, and with the subject looking in the forward direction with arms by their sides. Two visual conditions will be given: eyes-open (EO) and eyes-closed (EC). Each measurement will last for 60 seconds and will be repeated twice for each condition. A three-minute rest will be provided between measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.
2. Subject is male or female and is ≥ 65 and ≤ 85 years of age.
3. Subject has Body Mass Index (BMI) ≥ 20 but ≤ 32 kg/m2.
4. Subject is ambulatory and able to walk ≥ 25 meters without the use of an assistive device.
5. Subject has a serum 25-hydroxyvitamin D level ≥ 7.5 but ≤ 22.5 ng/ml (18.75 to 56.25 nmol/L) at screening.
6. Subject agrees to apply sunscreen (≥ SPF 30) on any exposed skin, when expecting an increase in exposure to sunlight (e.g. a planned holiday of more than eight days, a beach holiday or a holiday in the southern hemisphere, for the duration of the study).
7. Subject agrees not to use tanning beds for the duration of the study.
8. Subject agrees to refrain from starting any new exercise program, or weight loss program, for the duration of the study.
9. Subject is able to follow the protocol.

Exclusion Criteria:

1. Subject states they regularly consume supplemental vitamin D in the amount greater than the age-specific Institute Of Medicine daily recommended dietary allowance (600 IU or 15 µg for a subject ≥ 65 to ≤ 70 years of age; 800 IU or 20 µg for a subject > 70 years of age). Supplemental vitamin D includes standalone vitamin D supplements, vitamin D supplements with calcium, multi-vitamins, any medications containing vitamin D, and purposefully seeking sunlight when outdoors.
2. Subject states they have received vitamin D3 by injection within the last 3 months.
3. Subject is missing, or has had an amputation of, a limb.
4. For a subject who reports > 2 falls within the last year, or one fall within the last year with injury, study physician and study PI must approve participation in the study.
5. Subject states they have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
6. Subject states they have sarcoidosis, lymphoma, primary hyperparathyroidism, or any other disease that may enhance serum calcium concentration, as determined by the study physician.
7. Subject states they have had kidney stones within the last 3 years.
8. Subject states they have abnormal indices of calcium metabolism including hypercalcemia.
9. Subject states they have a granulomatous disease such as sarcoidosis, active chronic tuberculosis, and Wegener's granulomatosis.
10. Subject states they have been diagnosed with renal failure, renal insufficiency, or chronic kidney disease, or has received hemodialysis.
11. Subject states they have an active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix.
12. Subject states they have liver failure (decompensated chronic liver disease).
13. Subject has a stated history of a significant cardiovascular event (e.g., myocardial infarction, heart failure, or stroke) ≤ 3 months prior to screening visit.
14. Subject states they are currently diagnosed with, or has a history of severe dementia or delirium, eating disorder, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study dietary supplement consumption or compliance with study protocol procedures in the opinion of the principal investigator or study physician.
15. Subject reports having undergone major surgery, less than 6 weeks prior to enrollment in the study, or subject has planned inpatient surgery requiring 2 or more days of hospitalization during the entire study.
16. Subject states they have undergone hip replacement surgery within the last year.
17. Subject states they are currently being prescribed (by primary care physician or other health professional) medication that in the opinion of the study physician will have an effect on serum 25-hydroxyvitamin D levels (e.g., certain anticonvulsants, phenobarbital, carbamazepine, phenytoin).
18. Subject states they have been undergoing treatment within the last 2 years for epilepsy, and the treatment has an effect on serum 25-hydroxyvitamin D.
19. Subject states they have been prescribed within the last 2 years bisphosphonates or parathyroid hormone.
20. Subject states they cannot refrain from anabolic hormones or growth hormone, starting at screening and over the entire course of the study.
21. Subject reports alcohol intake as average of 3 or more servings per day (a serving defined as 4 oz wine, 12 oz beer, 1 oz spirits).
22. Subject states they have an allergy or intolerance to any ingredient in the study product.
23. Subject is deemed unsuitable for study based upon study physician assessment.
24. Subject is taking part in another clinical trial.
25. The use of fat absorption inhibiting products (e.g., prescription orlistat (Xenical), over the counter orlistat (Alli)) during the study.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dynamic Stability, change from baseline | 6 months
  Dynamic stability will be defined by the maximum Lyapunov exponent (maxLE), Floquet multiplier, or motor control timing, change from baseline. Dynamic stability, or walking stability, will be assessed with accelerometers while subjects are walking on a flat surface for about 60 seconds.

SECONDARY OUTCOMES:
Postural Stability, change from baseline | 6 months
  Postural stability will be measured in a still and standing subject, with foot placement standardized on a force plate, and with the subject looking in the forward direction with arms by their sides. Two visual conditions will be given: eyes-open (EO) and eyes-closed (EC). Each measurement will last for 60 seconds and will be repeated twice for each condition. A three minute rest will be provided between measurements.
Gait Speed, change from baseline | 6 months
  Participants will perform two bouts of walking at their usual pace along a flat surface. The two walks will be aggregated and average gait speed derived. Stride length, base width, sway will also be measured.
Handgrip Strength, change from baseline | 6 months
  Isometric handgrip strength will be measured with a hand dynamometer embedded with a strain gauge.
Timed get-up and go (TUG), change from baseline | 6 months
  Participants will be asked to stand from a seated position, walk 3 meters at their usual pace, turn around, walk back to the chair, and sit down.

OTHER OUTCOMES:
Blood Measures, change from baseline | 6 months
  Participants will be asked to provide blood for analysis of nutrient levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Glencroft Senior Living: Retirement Community in Arizona, Glendale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with Abbott Nutrition and DSM Nutritional Products, Inc.

REFERENCES:
- See also: Dietary Nutrient Information — https://www.nationalacademies.org/hmd/~/media/Files/Report%20Files/2010/Dietary-Reference-Intakes-for-Calcium-and-Vitamin-D/Vitamin%20D%20and%20Calcium%202010%20Report%20Brief.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-17): https://cdn.clinicaltrials.gov/large-docs/65/NCT02806765/Prot_SAP_000.pdf